CLINICAL TRIAL: NCT03842696
Title: A Phase 1/2 Multi-Center Trial of Vorinostat for Graft vs Host Disease Prevention in Children, Adolescents and Young Adults Undergoing Allogeneic Blood and Marrow Transplantation
Brief Title: Vorinostat for Graft vs Host Disease Prevention in Children, Adolescents and Young Adults Undergoing Allogeneic Blood and Marrow Transplantation
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UMCC 2018.081; HUM00147796 (Other: University of Michigan); HUM00186659 (Other: University of Michigan); UL1TR002240 (NIH)
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Diseases; Acute Leukemia in Remission; Chronic Myelogenous Leukemia - Chronic Phase; Chronic Myelogenous Leukemia, Accelerated Phase; Chronic Myelogenous Leukemia, Blastic Phase; Myelodysplastic Syndromes; Mantle Cell Lymphoma; Follicular Lymphoma; Diffuse Large B Cell Lymphoma; Non Hodgkin Lymphoma; Graft Vs Host Disease; Graft-versus-host-disease
Keywords: GVHD
MeSH Terms: conditions — Hematologic Diseases; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Myelodysplastic Syndromes; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Graft vs Host Disease | interventions — Vorinostat; Blood Specimen Collection; Tacrolimus; Cyclosporine; Methotrexate; Mycophenolic Acid; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vorinostat (Experimental)
  Interventions: Drug: Vorinostat; Procedure: Blood and Marrow Transplant (BMT); Drug: Tacrolimus (or cyclosporine); Drug: Methotrexate; Drug: Mycophenolate Mofetil (MMF); Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Vorinostat — * HLA-matched BMT recipients: Vorinostat 30, 45 or 60 mg/m2 BID (100 mg/m2 BID maximum) PO from 10 days prior to transplant (day -10), until day +30 post-transplant.
  * Haploidentical BMT recipients: Vorinostat 30, 45 or 60 mg/m2 BID (100 mg/m2 BID maximum) PO from 5 days after transplant (day +5), until day +30 post-transplant
Procedure: Blood and Marrow Transplant (BMT) — Undergo allogeneic BMT according to local site institutional practice.
Drug: Tacrolimus (or cyclosporine) — Tacrolimus (or cyclosporine if tacrolimus becomes in shortage during the study period) will begin on day -3. Intravenous or oral dosing is permitted.In the absence of GVHD, it is recommended that tacrolimus or cyclosporine tapering begin on day +100 post-transplant as per local site BMT program clinical practice guidelines. In the presence of GVHD, it is recommended that tacrolimus or cyclosporine be continued at therapeutic dosing.
Drug: Methotrexate — HLA-matched BMT recipients: Methotrexate will be used in combination with tacrolimus (or cyclosporine) for standard GVHD prophylaxis. It will be given at a dose of 5 mg/m2/dose once daily intravenously on days +1, +3, +6, and +11. Standard criteria for administration will be followed per local site institutional BMT program clinical practice guidelines.
Drug: Mycophenolate Mofetil (MMF) — Haploidentical BMT recipients: MMF will be used in combination with post-transplant cyclophosphamide and tacrolimus (or cyclosporine) for standard GVHD prophylaxis. MMF will start on day +5 and discontinue after the last dose on day +35 or may be continued if active GVHD is present. Given intravenously (preferred) or orally at a dose of 15 mg/kg/dose three times a day (based upon adjusted body weight) with the maximum total daily dose not to exceed 3 grams.
Drug: Cyclophosphamide — Haploidentical BMT recipients: Post-transplant cyclophosphamide (PT-Cy) will be used in combination with MMF and tacrolimus (or cyclosporine) for standard GVHD prophylaxis. PT-Cy (50 mg/kg/dose) given for two days, Days +3 and +4 after transplantation.

SUMMARY:
The purpose of this study is to determine the recommended phase 2 dose of the drug Vorinostat in children, adolescents and young adults following allogeneic blood or marrow transplant (BMT) and determine whether the addition of Vorinostat to the standard graft versus host disease (GVHD) prophylaxis will reduce the incidence of GVHD.

DETAILED DESCRIPTION:
All subjects will undergo allogeneic blood or marrow transplant (BMT) according to local site institutional practice. The preparative regimen will depend upon the subject's underlying disease, type of transplant, previous therapy and comorbidities. Stem cells can be from donors of bone marrow or peripheral blood stem cells.

ELIGIBILITY:
Inclusion Criteria:

* A prospective patient for allogeneic BMT for malignant hematologic conditions. A patient with history of CNS involvement is eligible if CNS disease is in remission at time of study consideration.
* The donor and recipient must have an HLA-match (8/8 HLA-A, -B, -C, and -DRB1) or haploidentical match (per protocol criteria). High resolution typing is required for all alleles.
* Diagnoses to be included:

  1. Acute Leukemia in remission. Remission is defined as the absence of blasts in the peripheral circulation at the time of enrollment, < 5% blasts in the bone marrow and absence of extramedullary disease including CNS involvement.
  2. Chronic Myeologenous Leukemia (CML) in first or subsequent chronic phase failing to respond (or intolerant) to at least two different tyrosine kinase inhibitors. CML in accelerated or blast phase (CML-AP/BP) are eligible without requirement to fail tyrosine kinase inhibitor therapy, but must be in remission at time of enrollment. Remission is defined as the absence of blasts in the peripheral circulation at the time of enrollment, <5% blasts in the bone marrow and absence of extramedullary disease including CNS involvement.
  3. Myelodysplastic syndrome (MDS) with intermediate or high-risk IPSS or equivalent IPSSR score with < 10% blasts in the bone marrow.
  4. Mature B Cell Malignancies (including Mantle Cell Lymphoma, Follicular Lymphoma. Diffuse Large B Cell Lymphoma, Non-Hodgkin Lymphoma not otherwise specified).Subjects should have extinguished standard of care options prior to being considered eligible for this trial
* Subjects aged 3 to 39 years
* Lansky/Karnofsky Performance Scale score of 70% or higher
* Life expectancy of greater than 6 months
* Subjects must have normal organ and marrow function (as defined in protocol)
* Ability to take oral medication and be willing to adhere to the vorinostat regimen
* For females of reproductive potential and men: The effects of vorinostat on the developing human fetus are unknown. For this reason and because histone deacetylase inhibitor agents as well as other therapeutic agents used in this trial (e.g., calcineurin inhibitor [tacrolimus or cyclosporine], methotrexate, mycophenolate, and cyclophosphamide) are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Women must continue using contraceptives for at least 6 months after the end of therapy and men must continue contraceptive use for 3 months after completion of vorinostat administration.
* Ability to understand and the willingness to sign a written informed consent document
* Stated willingness to comply with all study procedures and availability for the duration of the Study
* For the cognitive assessment and patient-reported QOL exploratory correlative portion of the study, subjects and caregiver must speak, read and understand English. Subjects who are too young to read must be able to understand and speak English, age-appropriately. Subjects who do not speak, read and understand English but satisfy all other inclusion criteria may still participate in the study but will not complete the cognitive and QOL portions.

Exclusion Criteria:

* Subjects who are not a candidate for an allogeneic BMT based on the current local site institutional BMT program clinical practice guidelines. Organ function criteria will be utilized per the current local site institutional BMT program clinical practice guidelines. There will be no restriction to study entry based on hematological parameters.
* Presence of anti-donor HLA antibodies (per protocol criteria).
* Subjects who are enrolled on another GVHD treatment or prevention trial.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Subjects still under therapy for presumed or proven infection are eligible provided there is clear evidence (radiographic findings and/or culture results) that the infection is well-controlled. Subjects under treatment for infection will be enrolled only after clearance from the PI.
* Pregnant women are excluded from this study because vorinostat is a histone deacetylase inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with vorinostat, breastfeeding should be discontinued if the mother is treated with vorinostat. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Subjects with evidence of HIV seropositivity and/or positive PCR assay, HTLV1/HTLV2 seropositivity. The safety of allogeneic HSCT is not yet well-established for this population.
* Subjects with evidence of Hepatitis B or Hepatitis C PCR positivity. Hepatitis reactivation following myelosuppressive therapy can lead to fatal complications.
* Subjects with a history of prolonged QTc syndrome.
* Subjects who have had prior treatment with a drug like vorinostat (i.e., valproic acid) within the last 30 days.
* Subjects with documented evidence of cognitive impairment prior to enrollment on this study (diagnosis of dementia, mild cognitive impairment, or other neurological illnesses that impacts cognition) are excluded from the cognitive assessment portion of the study only.

Ages: 3 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1 portion: Determine the recommended phase 2 dose (RP2D) of the drug Vorinostat in children, adolescents, and young adults following allogeneic blood or marrow transplant (BMT). | At day +100
  Real time assessment of safety (DLTs), and pharmacokinetic (PK) and pharmacodynamics/histone acetylation (PD) analysis in each dose cohort prior to escalation of dose. Dose de/escalation will be determined using the 3+3 up-or-down algorithm.
Phase 2 portion: Incidence of grade 2-4 acute GVHD within 100 days after transplant | At day +100
  Cumulative incidence will be determined using the proportional hazards method with a corresponding 95% confidence interval. GVHD severity will be determined clinically and graded by using the institutional BMT program clinical practice guidelines. (Pzrepiorka D, Weisdorf D, Martin P, et al. Consensus conference on acute GVHD grading. Bone Marrow Transplantation 1995; 15:825-8.)

SECONDARY OUTCOMES:
Incidence of Grade 3-4 acute GVHD within 100 days after transplant | At day +100
  Cumulative incidence will be determined using the proportional hazards method with a corresponding 95% confidence interval. GVHD severity will be determined clinically and graded by using the institutional BMT program clinical practice guidelines. (Pzrepiorka D, Weisdorf D, Martin P, et al. Consensus conference on acute GVHD grading. Bone Marrow Transplantation 1995; 15:825-8.)
Incidence of chronic GVHD | At 1 year
Incidence of relapse | At 1 year
  Determined using the proportional hazards method with a corresponding 95% confidence interval.
Overall Survival | At 1 year
  The Kaplan-Meier method will be used to estimate overall survival, measured from the date of transplantation to either death from any cause or end of follow-up.
Relapse-free Survival | At 1 year
GVHD-free relapse-free Survival | At 1 year
Number of participants with adverse events of grade 4 or higher that are probably or definitely related to vorinostat. | Up to day +100
  Graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Percentage of participants with engraftment failure | Up to 28 days post-transplant
  Engraftment failure will be defined as the inability to achieve an absolute neutrophil count (ANC) > 500/uL within 28 days post-transplant.
Percentage of participants for whom successful administration of at least 60% of the planned doses occurs between day -1 and day +30 post-transplant | Up to 30 days post-transplant
Maximum concentration (Cmax) of Vorinostat | At day +1
  Pharmacokinetic (PK) analysis will be performed using blood samples from subjects who have received at least one dose of vorinostat and for whom quantifiable PK samples are available. Pharmacokinetic variables will be summarized with descriptive statistics.
Area under the curve (AUC) of Vorinostat | At day +1
Clearance (CL) of Vorinostat | At day +1
Volume (V) of Vorinostat | At day +1

CONTACTS AND LOCATIONS:
Overall Officials: Sung W Choi, MD, MS, Principal Investigator — University of Michigan
Locations (7):
- United States (7):
  - University of Colorado, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No